CLINICAL TRIAL: NCT00590980
Title: The Vertebrobasilar Flow Evaluation and Risk of Transient Ischemic Attack and Stroke (VERiTAS) Study
Brief Title: Vertebrobasilar Flow Evaluation and Risk of Transient Ischemic Attack and Stroke (VERiTAS)
Acronym: VERiTAS
Status: Completed | Type: Observational
Sponsor: Sepideh Amin-Hanjani (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Sepideh Amin-Hanjani, Professor, Department of Neurosurgery, University of Illinois at Chicago, University of Illinois at Chicago
Organization: University of Illinois at Chicago (Other)
Other Study IDs: 2006-0599; 5R01NS059745 (NIH)
Record Dates: First submitted 2007-12-28; First posted 2008-01-11 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Vertebrobasilar Insufficiency; Ischemic Attack, Transient; Cerebrovascular Disorder; Brain Ischemia; Stroke
Keywords: Stroke; TIA (transient ischemic attack); Brain; Blood Flow; Quantitative magnetic resonance angiography (QMRA)
MeSH Terms: conditions — Vertebrobasilar Insufficiency; Ischemic Attack, Transient; Cerebrovascular Disorders; Brain Ischemia; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Patients with intracranial or extracranial vertebrobasilar occlusion or stenosis ≥ 50% presenting with vertebrobasilar distribution TIA or stroke.

SUMMARY:
Patients with blockage of the blood vessels that supply blood to the back of the brain, known as vertebrobasilar disease (VBD), are at risk of having a stroke or temporary symptoms of a stroke known as transient ischemic attack (TIA). The risk of repeated stroke associated with VBD may be affected by several risk factors, including the degree to which the blockage reduces the blood flow to the brain. Patients with VBD have different levels of blockage ranging from partial blockage to complete blockage, which can affect the blood flow to the brain by variable amounts. The purpose of this research is to determine if patients with symptomatic VBD who demonstrate low blood flow to the back of the brain on magnetic resonance (MR)imaging are at higher risk of developing another stroke or TIA than patients with normal blood flow.

DETAILED DESCRIPTION:
Approximately 700,000 strokes occur annually in the U.S. making it the third leading cause of death and the leading cause of permanent disability among adults. Over one third of strokes occur in the posterior circulation, the leading cause of which is vertebrobasilar occlusive disease secondary to atherosclerosis. Symptomatic vertebrobasilar disease (VBD) carries a high annual risk of stroke, averaging 10-15% per year despite medical therapy. This represents a potentially treatable high risk stroke etiology. Advances in endovascular angioplasty and stenting have created new treatment options, but these interventions carry significant risks, and the selection criteria for appropriate candidates remains uncertain. Determining predictors of stroke in this population is the first step toward identifying those high risk patients most suitable for consideration of intervention. Our preliminary studies suggest that the risk of stroke in VBD is strongly related to the extent to which intracranial blood flow is compromised.

The objective is to conduct a longitudinal study of patients with symptomatic VBD. Our central hypothesis is that patients with symptomatic VBD who demonstrate limitation of blood flow on quantitative magnetic resonance angiography (QMRA) are at higher risk of stroke.The primary aim of this proposal is to test the hypothesis that among patients with VBD, those with distal blood flow compromise are at higher risk of subsequent posterior circulation stroke than those with normal flow.

Secondary exploratory aims of the proposal are to determine:the correlation between large vessel flow measured by QMRA and tissue level perfusion measured by MR perfusion in the posterior circulation, and the predictive value of each; other predictive factors for stroke in this population; hemodynamic effects of varying degrees of vertebrobasilar stenosis; changes in hemodynamic status of patients on medical therapy over time; utility of QMRA as a non-invasive screening and monitoring tool in VBD.

The study is a prospective multi-center observational cohort study of patients with symptomatic angiographically confirmed vertebrobasilar atherostenosis (≥ 50%), or occlusion). Upon enrollment, patients will undergo hemodynamic assessment with noninvasive MR imaging (including QMRA and MR perfusion), the results of which will be kept blinded from treating physicians and the patients. Patients will be prospectively designated as demonstrating compromised or normal distal cerebral flow based upon an existing validated algorithm of individual posterior circulation vessel flow measurements. Baseline demographic, clinical and laboratory data will be gathered. Subsequently, patients will have monthly clinical follow-up and be re-imaged with QMRA at 6 month intervals for a minimum of 12 months. The primary endpoint will be stroke incidence in the vertebrobasilar territory at one year. Survival analysis methods, with censoring of patients not achieving endpoint at the end of the study period, will be used for comparison of patients with compromised versus normal blood flow.

The overall goal of the study is to define the population of patients with symptomatic VBD at highest risk of recurrent ischemic events. The information gained can significantly impact the selection criteria and likelihood for success of future clinical trials aimed at assessing the efficacy of endovascular or surgical interventions for the treatment of VBD. Moreover, the ability to define a low risk population in whom the risks of expensive invasive interventions would be unnecessary will have an equally important impact on the management of the disease both from a clinical and cost perspective. Data regarding the hemodynamic effects and changes over time of vertebrobasilar occlusive disease may also enhance our understanding of the basic pathophysiology and mechanisms of stroke in this morbid disease entity.

ELIGIBILITY:
Inclusion Criteria:

* Stroke or TIA in the vertebrobasilar territory
* Conventional or CT angiographic demonstration of ≥50% stenosis or occlusion of extracranial or intracranial vertebrobasilar artery
* Symptoms within 60 days of enrollment
* Age 18 and above
* Able to provide informed consent

Exclusion Criteria:

Neurologic criteria:

* Major disabling stroke prohibiting the ability to return for follow-up assessment
* Any neurological disease which would confound follow-up assessment

Medical criteria:

* Any severe co-morbidity condition with less than 12 month life expectancy
* Known cardiac disease associated with cardioembolic risk specifically atrial fibrillation, prosthetic valves, endocarditis, left atrial/ventricular thrombus, cardiomyopathy with EF<25%, cardiac myxoma
* Blood dyscrasias, specifically polycythemia vera, essential thrombocytosis, sickle cell disease

Disease criteria:

* Non-atherosclerotic disease vertebrobasilar disease including dissection, fibromuscular dysplasia, vasculitis, radiation induced vasculopathy
* Unilateral vertebral stenosis or occlusion

Patient criteria:

* Unable or unwilling to undergo MRI or cerebral angiography or CTA
* Pregnancy concurrent participation in an interventional trial for treatment of vertebrobasilar disease.
* Renal dysfunction will be exclusionary if it precludes angiography. No subjects will be excluded based upon gender, race, ethnic group, religion or socioeconomic status. Children will not be recruited as atherosclerotic VBD is a condition that affects adults primarily in later life and is not a disease that occurs or is relevant in children.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurology/Neurosurgery Clinic
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sepideh Amin-Hanjani, MD, Principal Investigator — University of Illinois, Department of Neurosurgery
Locations (6):
- United States (5):
  - University of California at Los Angeles - UCLA, Los Angeles, California
  - University of Illinois at Chicago, Chicago, Illinois
  - Jeffrey Kramer, MDSC at Mercy Hospital, Chicago, Illinois
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
- UHN-Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Amin-Hanjani S, Du X, Zhao M, Walsh K, Malisch TW, Charbel FT. Use of quantitative magnetic resonance angiography to stratify stroke risk in symptomatic vertebrobasilar disease. Stroke. 2005 Jun;36(6):1140-5. doi: 10.1161/01.STR.0000166195.63276.7c. Epub 2005 May 12. PMID 15890993
- [Background] Amin-Hanjani S, Rose-Finnell L, Richardson D, Ruland S, Pandey D, Thulborn KR, Liebeskind DS, Zipfel GJ, Elkind MS, Kramer J, Silver FL, Kasner SE, Caplan LR, Derdeyn CP, Gorelick PB, Charbel FT; VERiTAS Study Group. Vertebrobasilar Flow Evaluation and Risk of Transient Ischaemic Attack and Stroke study (VERiTAS): rationale and design. Int J Stroke. 2010 Dec;5(6):499-505. doi: 10.1111/j.1747-4949.2010.00528.x. PMID 21050408
- [Result] Amin-Hanjani S, Du X, Rose-Finnell L, Pandey DK, Richardson D, Thulborn KR, Elkind MS, Zipfel GJ, Liebeskind DS, Silver FL, Kasner SE, Aletich VA, Caplan LR, Derdeyn CP, Gorelick PB, Charbel FT; VERiTAS Study Group. Hemodynamic Features of Symptomatic Vertebrobasilar Disease. Stroke. 2015 Jul;46(7):1850-6. doi: 10.1161/STROKEAHA.115.009215. Epub 2015 May 14. PMID 25977279
- [Result] Amin-Hanjani S, Pandey DK, Rose-Finnell L, Du X, Richardson D, Thulborn KR, Elkind MS, Zipfel GJ, Liebeskind DS, Silver FL, Kasner SE, Aletich VA, Caplan LR, Derdeyn CP, Gorelick PB, Charbel FT; Vertebrobasilar Flow Evaluation and Risk of Transient Ischemic Attack and Stroke Study Group. Effect of Hemodynamics on Stroke Risk in Symptomatic Atherosclerotic Vertebrobasilar Occlusive Disease. JAMA Neurol. 2016 Feb;73(2):178-85. doi: 10.1001/jamaneurol.2015.3772. PMID 26720181
- [Result] Amin-Hanjani S, Turan TN, Du X, Pandey DK, Rose-Finnell L, Richardson D, Elkind MS, Zipfel GJ, Liebeskind DS, Silver FL, Kasner SE, Gorelick PB, Charbel FT, Derdeyn CP; VERiTAS Study Group. Higher Stroke Risk with Lower Blood Pressure in Hemodynamic Vertebrobasilar Disease: Analysis from the VERiTAS Study. J Stroke Cerebrovasc Dis. 2017 Feb;26(2):403-410. doi: 10.1016/j.jstrokecerebrovasdis.2016.09.044. Epub 2016 Oct 28. PMID 28029608
- [Derived] Amin-Hanjani S, See AP, Du X, Rose-Finnell L, Pandey DK, Chen YF, Elkind MSV, Zipfel GJ, Liebeskind DS, Silver FL, Kasner SE, Gorelick PB, Charbel FT, Derdeyn CP; VERiTAS Study Group. Natural History of Hemodynamics in Vertebrobasilar Disease: Temporal Changes in the VERiTAS Study Cohort. Stroke. 2020 Nov;51(11):3295-3301. doi: 10.1161/STROKEAHA.120.029909. Epub 2020 Oct 9. PMID 33032489
- [Derived] Amin-Hanjani S, Stapleton CJ, Du X, Rose-Finnell L, Pandey DK, Elkind MSV, Zipfel GJ, Liebeskind DS, Silver FL, Kasner SE, Caplan LR, Derdeyn CP, Gorelick PB, Charbel FT; VERiTAS Study Group. Hypoperfusion Symptoms Poorly Predict Hemodynamic Compromise and Stroke Risk in Vertebrobasilar Disease. Stroke. 2019 Feb;50(2):495-497. doi: 10.1161/STROKEAHA.118.023101. PMID 30580717
- [Derived] Esfahani DR, Pandey D, Du X, Rose-Finnell L, Charbel FT, Derdeyn CP, Amin-Hanjani S; VERiTAS Study Group. Cost-Effectiveness of Quantitative Magnetic Resonance Angiography Screening and Submaximal Angioplasty for Symptomatic Vertebrobasilar Disease. Stroke. 2018 Aug;49(8):1953-1959. doi: 10.1161/STROKEAHA.118.022339. PMID 30012817
- See also: VERiTAS Study website — http://veritas.neur.uic.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Patients with intracranial or extracranial vertebrobasilar occlusion or stenosis ≥ 50% presenting with vertebrobasilar distribution TIA or stroke.
Period: Overall Study
Arm/Group | All Study Participants
Started | 82
Completed | 72
Not Completed | 10
Not completed — Did not meet all inclusion criteria | 10

BASELINE CHARACTERISTICS:
Population: Analysis population consists of all participants meeting all inclusion/exclusion criteria
Groups:
- Study Participants: Patients with intracranial or extracranial vertebrobasilar occlusion or stenosis ≥ 50% presenting with vertebrobasilar distribution TIA or stroke.
Arm/Group | Study Participants
Number analyzed (Participants) | 72
Age, Continuous [Mean (Full Range); unit: years] | 65.6 [39 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 49
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Canada | 6
  United States | 66

OUTCOME MEASURES:

1. Primary Outcome: Fatal and Nonfatal Ischemic Stroke in the Vertebrobasilar Territory
Description: Definite fatal and nonfatal ischemic stroke in the vertebrobasilar territory
Time Frame: up to 27 months
Population: Study participants meeting all inclusion and exclusion criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 72
Participants | 72

ADVERSE EVENTS:
Time Frame: 1 year duration of participant participation.
Description: (AE) - related to the protocol MR imaging or angiogram (if the angiogram was performed as part of the study).
  (SAE) - related to the protocol MR imaging or angiogram results in the usual definition of an SAE.
Arm/Group | Observation
Serious Adverse Events (participants affected / at risk) | 0/82
Other Adverse Events (participants affected / at risk) | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2015-01-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT00590980/Prot_000.pdf